CLINICAL TRIAL: NCT01616407
Title: Effects of MDMA (Ecstasy) and Methylphenidate (Ritalin) on Social Cognition
Brief Title: Effects of MDMA and Methylphenidate on Social Cognition
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 382/11; 2012DR1018 (Other: Swissmedic)
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Social Cognition
Keywords: Effects of psychostimulants on emotion recognition and empathy
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDMA, methylphenidate, placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but three treatment conditions in the same subject.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — 75 mg per os, single dose
  Other Names: - MDMA; - ecstasy
Drug: Methylphenidate — 40 mg per os, single dose
  Other Names: - Ritalin; - Concerta
Drug: Placebo — capsules identical to MDMA or methylphenidate but containing no active drug

SUMMARY:
The purpose of this study is to assess and compare the effects of a single dose of 3,4-methylenedioxymethamphetamine (MDMA)and methylphenidate (MPH) on emotional and social cognition in healthy subjects. The investigators hypothesize that MDMA enhances affective perception for positive and impairs perception for negative emotional stimuli compared to placebo or MPH.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except THC-containing products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Effects on social cognition (emotion recognition and empathy) | 7 hours

SECONDARY OUTCOMES:
Blood pressure (mmHg) and heart rate (beats per min) | 7 hours
Subjective effects | 7 hours
  subjective effects are repetitively assessed by standardized questionnaires
Neuroendocrine plasma levels | 7 hours
  neuroendocrine parameters assessed: prolactin, cortisol, epinephrine, norepinephrine, oxytocin, pro-vasopressin, vasopressin, estrogene,and progesterone
Drug plasma concentration | 7 hours
  The plasma concentration of MDMA and MPH is repetitively assessed.

OTHER OUTCOMES:
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Schmid Y, Hysek CM, Simmler LD, Crockett MJ, Quednow BB, Liechti ME. Differential effects of MDMA and methylphenidate on social cognition. J Psychopharmacol. 2014 Sep;28(9):847-56. doi: 10.1177/0269881114542454. Epub 2014 Jul 22. PMID 25052243